CLINICAL TRIAL: NCT06177288
Title: A Prospective, Single-arm Clinical Study on the Efficacy and Safety of DEBIRI Combined With Systemic Chemotherapy and Bevacizumab for Unresectable Colorectal Cancer With Liver Metastases
Brief Title: DEBIRI Combined With Chemotherapy and Bevacizumab in the Treatment of Unresectable Colorectal Cancer Liver Metastases
Acronym: DEBIRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Chief Physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-331R
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DEBIRI (Experimental): After dissolving 100 mg of irinotecan in water for injection or 4 ml of 5% glucose water, use 2 mL of 70 μm uniform particle size microspheres for loading and adsorption for 5 minutes. Then mixed with non-plasma contrast agent to embolize the tumor feeding artery.
  Interventions: Combination Product: DEBIRI Combined With Chemotherapy and Bevacizumab

INTERVENTIONS:
Combination Product: DEBIRI Combined With Chemotherapy and Bevacizumab — After dissolving 100 mg of irinotecan in water for injection or 4ml of 5% glucose water.use 2mL of 70μm uniform particle size microspheres for loading and adsorption for 5minutes. Then mixed with non-plasma contrast agent to embolize the tumor feeding artery.

SUMMARY:
To study the efficacy and safety of embolization therapy with uniform particle size drug-eluting beads loaded with irinotecan (DEBIRI) in patients with unresectable colorectal cancer liver metastases.

DETAILED DESCRIPTION:
Colorectal cancer is the second most common malignant tumor and the fifth cause of cancer death in my country, and its incidence rate is increasing year by year. The liver is the main target organ for hematogenous metastasis of colorectal cancer and the main cause of death in patients with colorectal cancer. About 15% to 25% of patients with colorectal cancer have liver metastases when diagnosed, and another 15% to 25% of patients will develop liver metastases after radical resection of the primary colorectal cancer site. The vast majority (80%) %~90%) of liver metastases cannot be curatively resected initially. The median survival of patients with untreated liver metastases is only 6.9 months, and the 5-year survival rate of patients with unresectable liver metastases is less than 5%. The median survival time of patients who have completely resected liver metastases or reached a state of no evidence of disease is 35 months, and the 5-year survival rate can reach 30% to 57%.

For patients with unresectable colorectal cancer liver metastases, the first-line treatment option recommended by the guidelines is multi-agent chemotherapy with or without targeted therapy.

Currently, there are limited clinical studies on the use of uniform particle size drug-loaded microspheres combined with chemotherapy drugs and targeted drugs to treat unresectable colorectal cancer liver metastases. Based on this, a single-arm, prospective study is planned to be carried out, using conversion resection rate as the main efficacy indicator, to explore the efficacy of embolization therapy with uniform particle size drug-loaded microspheres loaded with irinotecan combined with systemic chemotherapy and bevacizumab versus systemic chemotherapy combined The efficacy and safety of bevacizumab in the treatment of patients with unresectable colorectal cancer liver metastases provide a more reliable basis for clinical treatment in this field.

ELIGIBILITY:
Inclusion Criteria:

* 1: Age 18-75, no gender limit
* 2: Colorectal cancer liver metastasis diagnosed by histopathology/imaging or clinically (refer to the "Guidelines for the Diagnosis and Comprehensive Treatment of Colorectal Cancer Liver Metastasis" 2023 Edition)
* 3: The liver is the main target organ for distant metastasis (defined as ≥80% tumor burden limited to the liver)
* 4: The liver metastasis is determined to be initially unresectable after discussion by the MDT of the research center
* 5: There is at least one measurable liver metastasis, and the tumor diameter is >1cm (mRECIST assessment)
* 6: Liver metastases without interventional treatment (TACE, ablation, iodine particle therapy, etc.)
* 7: The tumor accounts for less than 60% of the total liver
* 8: The primary tumor is removed or still exists
* 9: Have not received anti-tumor treatment in the past or it has been more than 1 year since the last anti-tumor treatment
* 10: Expected survival >3 months
* 11: Liver function Child-Pugh class A or B
* 12: ECOG ≤2 points
* 13: Adequate renal function (creatinine ≤ 2.0mg/dl)
* 14: Women of childbearing age and men of childbearing potential voluntarily take appropriate contraceptive measures during treatment
* 15: Understand and sign the informed consent form

Exclusion Criteria:

* 1: Combined with other malignant tumors, except for cervical cancer in situ or cutaneous squamous cell carcinoma that has been fully treated, or basal cell carcinoma of the skin that has been basically controlled, except for colorectal cancer
* 2: There are any contraindications to TACE treatment
* 3: Patients eligible for radical treatment (surgery or ablation)
* 4: Any contraindications to irinotecan: chronic inflammatory bowel disease and/or intestinal obstruction
* 5: history of severe allergic reaction to irinotecan hydrochloride trihydrate, lactic acid or lactic acid and mannitol or the excipients in this product
* 6: Severe bone marrow failure
* 7: history of Gilbert syndrome (no specific testing required)
* 8: Those with brain metastases or a history of uncontrollable mental illness or severe intellectual or cognitive impairment
* 9: Severe active infection requiring intravenous antibiotic treatment occurs during the screening period
* 10: Active bleeding or abnormal coagulation function (PT> 16s, APTT> 43s, INR> 1.5 x ULN), or bleeding tendency or undergoing thrombolytic treatment
* 11: Patients with serious heart, brain, liver, and kidney system diseases
* 12: Unstable angina, angioplasty, stent placement or myocardial infarction within 6 months
* 13: Pregnant or lactating women, and those who are of childbearing potential but refuse to take contraceptive measures
* 14: Those who are allergic to experimental drugs
* 15: Patients who cannot comply with the trial protocol or cannot cooperate with follow-up visits
* 16: Those who the researcher believes are not suitable to participate in this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
converted resection rate | 1, 3, 6 months after surgery
  Discussed and determined by the MDT of the research center.

SECONDARY OUTCOMES:
Actual R0 resection rate | 1, 3, 6 months after surgery
  Postoperative pathological examination.No cancer cells can be found at the resection margin of the postoperative specimen under a microscope. There are no cancer cells remaining either to the naked eye or under a microscope, and the lesion has been completely removed.
Progression Free Survival | 1, 3, 6 months after surgery
  Time from initiation of treatment to tumor progression or death from any cause, whichever occurs first
Recurrence-free survival | 1, 3, 6 months after surgery
  Time from date of curative surgery to recurrence or death
Adverse events | 1, 3, 6 months after surgery
  Adverse medical events that occur to subjects during clinical trials

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Jianmin, Ph.D, Principal Investigator — Fudan University
Locations (1):
- Zhongshan hospital, Fudan university, Shanghai, China